CLINICAL TRIAL: NCT03038646
Title: A Phase 1, Open-Label, Randomised, 3-Treatment, 3-Period, Single-Dose, Crossover Study in Healthy Subjects to Compare the Pharmacokinetic Properties of Modified Release (MR) Formulations of MIN-101 Followed by Food Effect Testing of a Selected Formulation
Brief Title: A Pharmacokinetic Study of Modified Release (MR) Formulations of MIN-101 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minerva Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MIN-101C06
Record Dates: First submitted 2017-01-10; First posted 2017-02-01 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Food Effect
MeSH Terms: interventions — roluperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Regimen A (Experimental): 32 mg MIN-101 of the current modified-release formulation (comparator) identified as MR-32 formulation administered in the fasted state
  Interventions: Drug: MIN-101
- Regimen B (Experimental): 32 mg MIN-101 MR administered in the fasted state
  Interventions: Drug: MIN-101
- Regimen C (Experimental): 32 mg MIN-101 MR administered in the fasted state
  Interventions: Drug: MIN-101
- Part 2 selected dose (Experimental): 32 mg MIN-101 of MR administered in the fed state
  Interventions: Drug: MIN-101

INTERVENTIONS:
Drug: MIN-101

SUMMARY:
* To evaluate the pharmacokinetic (PK) profiles of MIN-l0l following administration of modified release (MR) formulations of MIN-l0l in healthy male and female subjects
* To select 1 MR formulation for use in fed state
* To evaluate the effect of food on the bioavailability of MIN-l0l selected MR formulation

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed CYP 2D6 extensive metaboliser genotype
2. Subject has given voluntary written informed consent before performance of any study related procedure
3. Must be 18 to 45 years of age, inclusive
4. Subject must be a healthy male or female as indicated by the protocol
5. Agree to abstain from all medication (except for allowed birth control for 21 days before the first dose with MIN-101
6. Subject agrees to use the methods of birth control as outlined in the protocol
7. Must be willing and able to communicate and participate in the whole study.
8. Willing to eat all the food supplied throughout the study.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal disease, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic or psychiatric disease or any other condition which, in the opinion of the principle investigator, would jeopardize the safety of the subject or impact the validity of the study results
2. Acute diarrhoea or constipation in the 7 days before the predicted first study day.
3. Subject has donated blood within 90 days or plasma within 30 days of study dosing
4. Regular alcohol consumption in males> 21 units per week and Females > 14 units per week (1 Unit = 1/2 pint beer, 25 mL of 40or a 125 mL glass of wine)
5. Subject has a borderline or long QTc Fridericia interval as defined by screening readings of >430 msec for males and >440 for females or a personal or familial history of long QT syndrome
6. Subject has participated in a clinical trial within 90 days prior to study initiation
7. Females who are pregnant or breast feeding
8. Subject has used any prescription medication or over-the-counter (OTC) medication, including vitamin supplements, within 21 days prior to day l
9. Subject has been treated with any known P450 206 or 3A4 enzymes altering drugs within 30 days prior to the study
10. Subject has smoked or used nicotine products within 2 months prior to or during the study
11. Subject has sought advice from or been referred to a GP or counsellor for abuse or misuse of alcohol, non-medical drugs, medicinal drugs or other substance abuse, e.g. solvents
12. Subject has a positive blood screen for HIV, Hepatitis B surface antigen (HBsAg), and Hepatitis C Antibody
13. Any current or previous use of drugs such as opiates, cocaine, ecstasy, or intravenous amphetamines and/or a positive urine screen for alcohol or drugs of abuse. Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs-of-abuse test and have been abstinent from cannabis use for at least 3 months
14. Subject has a current uncontrolled inter-current illness (i.e., active infection) or has had a clinically significant illness within the last 30 days prior to Day 1
15. Subject has had major surgery within 28 days of study entry, or 12 months prior to study for gastrointestinal surgery.
16. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Part 1: Plasma PK parameter, Cmax | from predose up to 72 hours post dose: Blood samples for MIN-101 will be collected at time 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 48, 60, and 72 hours post-dose on Day 1 of all periods.
  To estimate the relative bioavailability of MIN-l0l following MIN-101 administration. Plasma samples will be analyzed for MIN-101 and its metabolites using a validated LC-MS/MS method
Part 1: Plasma PK parameter, Tmax | from predose up to 72 hours post dose
Part 1: Plasma PK parameter, Tlag | from predose up to 72 hours post dose
Part 1: Plasma PK parameter,partial AUC (e.g., AUC12, AUC24), AUClast, AUC∞ | from predose up to 72 hours post dose
Part 1: Plasma PK parameter, λz and t1/2 | from predose up to 72 hours post dose
Part 2: Plasma PK parameter, Cmax | from predose up to 72 hours post dose: Blood samples for MIN-101 will be collected at time 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 10, 12, 14, 16, 20, 24, 28, 32, 36, 48, 60, and 72 hours post-dose on Day 1 of all periods.
  To estimate the relative bioavailability of MIN-101 and its main metabolites following the administration of the selected modified release formulation in different food conditions (fasted or fed state).
Part 2: Plasma PK parameter, Tmax | from predose up to 72 hours post dose
Part 2: Plasma PK parameter, Tlag | from predose up to 72 hours post dose
Part 2: Plasma PK parameter, λz and t1/2 | from predose up to 72 hours post dose

SECONDARY OUTCOMES:
Part 1: QTcF changes from baseline | from predose up to 72 hours post dose
  The effect of coincidentally measured (time-matched) plasma concentrations of MIN-l0l on QTcF changes from Baseline.
Part 1: Safety (AE reporting, safety laboratory parameters analysis, vital signs and 12 lead ECG assessments) | 2 months 16 days
  Safety will be assessed through AE reporting, safety laboratory parameters analysis, vital signs and 12 lead ECG assessments
Part 2: Safety (AE reporting, safety laboratory parameters analysis, vital signs and 12 lead ECG assessments) | 2 months 16 days
  Safety will be assessed through AE reporting, safety laboratory parameters analysis, vital signs and 12 lead ECG assessments

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jabbari, MD, Principal Investigator — BioKinetic Europe Ltd
Locations (1):
- Biokinetic Europe, Belfast, Ireland

IPD SHARING:
Plan to Share IPD: No